CLINICAL TRIAL: NCT01037140
Title: Effects of Vitamin D Supplementation in Vitamin D Deficient Obese Subject.
Brief Title: Effects of Vitamin D Supplementation in Obesity
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2008-005581-31
Record Dates: First submitted 2009-12-08; First posted 2009-12-21 (Estimated); Last update posted 2012-08-02 (Estimated); Status verified 2012-08

CONDITIONS: Vitamin D Deficiency; Obesity
MeSH Terms: conditions — Vitamin D Deficiency; Obesity | interventions — Cholecalciferol; Vitamin D

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- cholecalciferol (Active Comparator)
  Interventions: Drug: Cholecalciferol
- placebo (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Cholecalciferol — oral cholecalciferol tablets of 175 micrograms daily for 6 months
  Other Names: vitamin D
  Arms: cholecalciferol
Drug: placebo — oral placebo tablets similar to active comparator
  Arms: placebo

SUMMARY:
Obesity is an increasing health problem with numerous metabolic complications. Vitamin D deficiency is common in obesity, and in epidemiological studies vitamin D deficiency has been linked to metabolic complications, such as type 2 diabetes, insulin resistance and cardiovascular disease, as well as myopathy, osteoporosis and depression. In obesity, a low grade inflammation is present in the fat tissue, thereby releasing inflammatory molecules to the blood stream. In cell line studies as well as small clinical studies vitamin D has been shown to have the ability to reduce inflammation and cell growth.

In the present study the investigators wish to investigate the effect of vitamin D on fat-, muscle and bone metabolism. 30 healthy obese subjects will be treated with cholecalciferol 175 micrograms daily for 6 months and will be compared with 30 healthy obese subjects treated with placebo.

The investigators hypothesize that restoring vitamin D levels in vitamin D deficient obese subject will reduce inflammation and thereby reduce obesity-related complications.

The effect will be evaluated as follows:

* Levels of circulating inflammatory markers will be examined in blood samples collected prior to and after treatment.
* Effects on fat- and muscle metabolism will be evaluated in fat- and muscle samples taken before and after treatment.
* Effects on fat distribution will be evaluated by MRI scan before and after treatment.
* Effects on insulin sensitivity will be evaluated by hyperinsulinaemic euglycaemic clamp performed on a subgroup of subjects with impaired fasting glucose.
* Effects on bone marrow density will be evaluated by DEXA scans before and after treatment.
* Effects on quality of life and depression score will be evaluated by questionnaires used before and after treatment.

ELIGIBILITY:
Inclusion Criteria:

* Healthy obese (BMI 30 - 45 kg/m2)
* 25(OH) vitamin D < 50 nmol/l

Exclusion Criteria:

* Diabetes,
* Pregnancy or non-safe contraception,
* Vitamin D treatment within 3 months,
* Hypercalcaemia, renal failure,
* Liver failure, non eligibility for MRI-scan,
* Severe osteomalacia,
* Allergy towards study drug

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 55 (Actual)
Dates: Start 2010-01; Primary Completion 2011-12 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Effect on circulating inflammatory markers | 6 months

SECONDARY OUTCOMES:
change in fat distribution | 6 months
change in insulin sensitivity | 6 months
change in bone mineral density | 6 months
change in quality of life | 6 months
change in depression score | 6 months
change in muscle function | 6 months
change in fat- and muscle metabolism | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Louise Wamberg, Dr., Principal Investigator — Aarhus University Hospital
Locations (1):
- Dept. of Endocrinology and Metabolism, Aarhus University Hospital, Aarhus, Denmark

REFERENCES:
- [Derived] Bislev LS, Wamberg L, Rolighed L, Grove-Laugesen D, Rejnmark L. Effect of Daily Vitamin D3 Supplementation on Muscle Health: An Individual Participant Meta-analysis. J Clin Endocrinol Metab. 2022 Apr 19;107(5):1317-1327. doi: 10.1210/clinem/dgac004. PMID 35018442